CLINICAL TRIAL: NCT00869830
Title: The Effectiveness of Biofeedback Treatment in Constipated Patients With Idiopathic Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Seung-Jae, Myung, Assistant Professor, Asan Digestive Disease Research Institute, Department of Internal Medicine, University of Ulsan College of Medicine, Asan Medical Center, Seoul, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFT in IPD
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Idiopathic Parkinson's Disease; Constipation
Keywords: Biofeedback; constipation; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Constipation | interventions — Biofeedback, Psychology; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- biofeedback (Experimental)
  Interventions: Other: biofeedback therapy

INTERVENTIONS:
Other: biofeedback therapy — biofeedback therapy was applied using the surface electromyography (EMG) method with a perianal sensor (Perry, Elan, SRS Medical Systems, Redmond, WA, USA) and biofeedback PC equipment (Orion, Platinum, SRS Medical Systems, Inc., Redmond, WA, USA).
  Other Names: perianal sensor (Perry, Elan, SRS Medical Systems, Redmond, WA, USA); biofeedback PC equipment (Orion, Platinum, SRS Medical Systems, Inc., Redmond, WA, USA).

SUMMARY:
The aims of the investigators' study are to characterize the nature of constipation in idiopathic Parkinson's disease (IPD) and to evaluate the usefulness of biofeedback therapy in constipated IPD patients.

DETAILED DESCRIPTION:
The medical treatment of idiopathic Parkinson's disease (IPD) alleviates constipation symptoms due to the restoration of autonomic dysfunction. However, additional laxatives are usually needed in these patients. Other suppository treatments included stool softeners, dopamine-receptor agonists, botulinum toxins, and prokinetic medications such as tegaserod. Biofeedback therapy (BFT) has been the gold standard for functional constipation with dyssynergic defecation or rectal hyposensitivity. However, researchers have not tried to evaluate its usefulness in constipated IPD patients up to now. The aims of our study are to characterize the nature of constipation in IPD and to evaluate the usefulness of BFT in constipated IPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease

Exclusion Criteria:

* Secondary Parkinson's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of biofeedback therapy in Parkinson's disease | usually six sessions per one biofeedback for 3 months

SECONDARY OUTCOMES:
to evaluate the constipation type in Parkinson's disease | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kee Wook Jung, M.D., Principal Investigator — Asan Digestive Disease Research Institute, Department of Internal Medicine, University of Ulsan College of Medicine, Asan Medical Center, Seoul, Korea
Locations (1):
- Seung-Jae, Myung, Seoul, Seoul, South Korea